CLINICAL TRIAL: NCT04406350
Title: Feasibility Study of Isoxic/Normocapnic End-tidal Gas Control to Decrease Incidence of Postoperative Delirium (POD) During Anesthetic Management
Brief Title: Tight End-tidal Gas Control During Anesthesia to Decrease Postoperative Delirium Anesthetic Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOC2019-6
Record Dates: First submitted 2020-02-19; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-02

CONDITIONS: Post-Operative Confusion; Delirium; Anesthesia Complication
Keywords: anesthesia; post-operative delirium; MRI; BOLD imaging; psychometric testing
MeSH Terms: conditions — Delirium; Emergence Delirium

STUDY DESIGN:
Intervention Model Description: A pilot study to determine the feasibility of tight control of end-tidal respiratory gases during the conduct of anesthesia in major surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group - MRI CO2 and O2 stress test (Experimental): Pilot Study of Feasibility of tight control of end-tidal respiratory gases during conduct of anesthesia
  Interventions: Procedure: Intraoperative tight control of respiratory end-tidal gases

INTERVENTIONS:
Procedure: Intraoperative tight control of respiratory end-tidal gases — Control of ET CO2 and ET O2 during conduct of anesthesia.

SUMMARY:
Respiratory end-tidal gas control is a fundamental of anesthetic management. The range of end-tidal (ET) O2 and CO2 during the conduct of anesthesia is far outside that found in the awake state. Recent work has indicated that alterations in end-tidal gases may influence the incidence of postoperative delirium (POD). This study will examine the feasibility of tight end-tidal gas control during anesthesia to decrease the incidence of POD.

DETAILED DESCRIPTION:
A. Background and Rationale:

Although respiratory end-tidal gas control is a fundamental principle of anesthetic management, the range of end-tidal (ET) O2 and CO2 typically seen during the conduct of anesthesia can significantly deviate from the awake baseline state, but has not been considered as a potential contributor to POD in previous investigations. Periods of both hypocapnia during mechanical ventilation and hypercapnia during the reestablishment of spontaneous ventilation are common. The use of 100% oxygen during anesthesia induction and emergence and maintenance of anesthesia with O2 concentrations of 50% are typical. The effects of these alterations in respiratory gases have significant effects on cerebral blood flow and oxygenation, which may be implicated in cognitive dysfunction. The investigators plan to examine the effects of controlled alterations in ET O2 and CO2 during anaesthesia and surgery on the incidence of POD.

B. Hypothesis and Study Objectives:

The investigators advance the hypothesis that ET respiratory gas control is a critical management consideration during anaesthesia; a much more important consideration than previously thought. Older patients appear to be at greater risk of 'intracranial steal' of regional CBF with alterations in CO2 and O2. The investigators previous study confirms an association between CO2 management and POD. Prior MR imaging suggests that a combination of hyperoxia and hypocapnia may be particularly worrisome, a very common situation during anesthesia. The investigators suggest that anesthetic management may be optimized for cerebral health by attempting to maintain respiratory gases at or near the patient baseline values to stabilize CBF during the conduct of anesthesia. An exception occurs during neurosurgical procedures where deliberate alterations to lower ET CO2 may be required. The marked CBF fluctuations as seen with controlled ET gas manipulation in our prior work imply that such CBF changes can occur under anesthesia where similar changes in ET gases routinely occur. The investigators propose that such large alterations in CBF and oxygenation may be a contributing factor to the development of POD in susceptible individuals. Here is proposed a feasibility trial of rigorous maintenance of ET gases at a patient's own baseline to study if such management has an influence on the incidence of POD.

C. Methodology: Summarize study location (facility), eligibility criteria, details regarding recruitment, consent, and randomization, interventions(s), covariates, data sources as applicable.

Twelve patients undergoing high-risk surgeries requiring a post-operative stay will be approached to participate in the study through the Pre-Anesthesia Clinic (PAC) at the HSC. Witnessed informed consent will be obtained from each patient. Exclusion criteria will include simultaneous planned carotid endarterectomy, carotid stenosis-if previously documented, planned neurosurgical procedures, contraindications to MRI including claustrophobia, expected one-lung anesthesia, and known chronic obstructive lung disease with CO2 retention. Patients will be seen pre-operatively in the week prior to surgery for comprehensive neuropsychological testing followed immediately by the MRI BOLD CO2 and O2 stress test. A trained psychometrist will administer a battery of neuropsychological tests over the span of approximately 1 hour. Subsequently, the MRI BOLD stress testing will be undertaken. Patients will undergo their surgery with no alterations to their anesthesia management except ET CO2 at ±2.5 mm Hg of baseline and FiO2 at 0.3, post induction This will be correlated to arterial blood gases to maintain arterial O2 at 125±25 mm Hg. Following surgery, trained personnel blinded to pre-operative performance on all assessments will conduct daily POD assessments for up to 5 post-operative days including day 0 (day of surgery). Patients will be contacted via phone at least 1 month post-operatively and asked about their cognition since their surgery.

Diathesis Assessments- Pre-operative Psychiatric and Neuropsychological Assessments: Upon initial recruitment in PAC, patients will complete the validated Patient Health Questionnaire (PHQ-9) to assess depressive symptoms and the Generalized Anxiety Disorder Scale (GAD-7) to assess anxiety symptoms, and self-report on psychiatric disorder diagnoses previously made by health professionals. For neuropsychological testing, attention will be assessed using Trails A and Weschler Adult Intelligence Scale (WAIS)-IV Digit Span; information processing speed using WAIS-IV Digit Symbol Coding; verbal memory using Hopkins Verbal Learning Test-Revised; visual construction, planning and organization using Rey's Complex Figure (copy trial); visual memory using Rey's Complex Figure (immediate recall trial); executive functioning/processing speed using Trails B and Delis-Kaplan Executive Function System (DKEFS) Color Word Interference; verbal and semantic fluency using F-A-S and Animal Fluency; spatial skills using CLOX I (free draw) and II (copy); and global cognitive and mental status using the Mini-Mental Status Examination (MMSE).

Pre-operative Neuroimaging and CO2 and O2 Stress Test: The CO2 and O2 stress test will be conducted during neuroimaging where all participants had model-based prospective end-tidal (MPET) CO2 targeting achieved by precise delivery of CO2 and O2 at a fixed concentration using a sequential breathing circuit regulated by a computerized gas-blender (RespirAct™, Thornhill Research Inc., Toronto, ON). This device allows precisemanipulation of end tidal CO2 levels and determines patient baseline ET CO2 values under isoxic conditions and precise end tidal O2 under isocapnic conditions. All MR images will be acquired using a Siemens Verio 3.0T MR scanner with a 12-channel phased-array head coil.

Stressor Assessments - Intra-operative Assessments: An arterial cannula will be inserted to monitor blood pressure and for serial ABG determination. A baseline ABG will be drawn to determine resting arterial CO2 and O2 on room air. These measures will determine the target points for end-tidal gas values for the duration of the anesthesia. All patients will receive a general anesthetic-either sevoflurane or desflurane as volatile agent in air:O2. Immediately following induction FiO2 will be set at 0.3 and end-tidal CO2 determined based on the value of the arterial CO2 and the recorded difference in the A-a CO2 gradient as measured from simultaneous end-tidal CO2. For the duration of the anesthetic, including emergence the end-tidal CO2 will be adjusted to no greater than ±2.5 mmHg from the determined value. If end-tidal O2 is satisfactory and pulse oximetry is above 98% then the FiO2 will be unchanged. If FiO2 is greater than 0.5 for greater than 15 minutes at any time the study will be terminated with patient management at the discretion of the attending anesthesiologist. Hemodynamics, end-tidal gas tensions (O2, CO2 and anesthetic vapour) will be recorded at 1 hz using a data acquisition system and stored on a laptop computer. At the end of their surgical procedure all patients will be initially monitored in the recovery room and then transferred either to the surgical intensive care, or the inpatient surgical wards. The data stream will be processed, collated with Excel, and transferred to SPSS for analysis.

Post-operative Assessment for Delirium: A trained blinded interviewer will conduct the CAM-S, a structured 10-15 min clinical interview, to assess the presence and severity of POD. The total severity score will be based on a sum score that could range from 0 through 19. The investigators will report the peak post-operative severity score for each patient throughout their inpatient stay and the average severity score up to 5 post-operative days (unless discharged prior to 5 days). Subthreshold delirium (ST-POD) will be defined as those not meeting full criteria but displaying elevated severity scores (≥5) on the POD severity long form on at least 1 post-operative day.

Statistical Analyses: BOLD imaging will be processed as 1st and 2nd level analysis by SPM. Second level analysis has defined cut-points for abnormal image patterns for voxel counts based on an adult atlas of normal controls developed at this institution. Perioperative data will be analyzed using SPSS. Bivariate correlations will examine the relationship between cognitive summary scores and psychiatric severity scores as indicated by PHQ-9 and GAD-7 with continuous severity POD measures. If significant results are indicated, a bivariate linear regression model will be conducted followed by a model controlling for age, education, sex and pre-operative baseline POD severity. The investigators will also conduct analyses of variance to examine mean score differences across primary diathesis and stress factors among those classified as non-POD, ST-POD, and full POD.

D. Primary Outcome:

Feasibility study of ease of end-tidal gas control of CO2 and O2 to defined targets intraoperatively.

E. Secondary Outcomes:

Correlations of POD using this management approach with other outcome markers in our stress-diathesis model. Ease of maintenance of this anesthetic approach. Assessment of adverse outcomes.

F. Feasibility: Justify the sample size with a power analysis. If a power analysis was not done, state why. For prospective studies, discuss expected duration of study of terms of expected number of eligible participants, recruitment rate and attrition rate. For retrospective studies, relate the sample size to the available data.

All technical aspects of this proposed study have been established, including the comprehensive psychometric testing, MR imaging and high fidelity data acquisition in the operating room. A knowledgeable team capable of carrying out this feasibility study is in place at HSC. This proposed study is underpowered to definitively make an assessment of the merits of controlled end-tidal gas control. This study will examine the feasibility of the approach in 12 patients. Based on a 50% reduction of POD (perhaps optimistic, at an α of 0.05 and a β of 0.80 the investigators envision requiring 136 patients to truly assess the merits of the approach when compared to a standardly management group. This is within the feasibility of a single centre but such an estimation may be overly zealous.

G. State the expected results:

The investigators expect to demonstrate a decrease in the incidence of POD in this feasibility study at 50% of that seen in our prior study (25% incidence for full POD). Outcome data from this study will be used to establish a formal power analysis of POD incidence to permit a more formal and comprehensive RCT based on PACT participation.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* elective major surgery requiring a minimum stay of 2 days postoperatively
* no contraindication to MRI

Exclusion Criteria:

* unable to provide informed consent
* CO2 retention with Chronic Obstructive Pulmonary Disease (COPD)
* active congestive heart failure (CHF)
* unable to participate adequately in delirium screening including those who are blind, deaf, illiterate or not fluent English or French
* prior episode of intraoperative awareness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-operative delirium | 5 days
  Incidence of delirium will be assessed in the Pilot Study Group as measured by the number of positive Confusion Assessment Method (CAM) and CAM-S or CAM for intensive care unit (CAM-ICU) scores, coupled with Chart Review.

SECONDARY OUTCOMES:
Length of Hospital stay | Time (days) from admission to discharge from hospital (or through study completion at one year)
  Length of hospital stay (days) will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mutch WAC, El-Gabalawy R, Girling L, Kilborn K, Jacobsohn E. End-Tidal Hypocapnia Under Anesthesia Predicts Postoperative Delirium. Front Neurol. 2018 Aug 17;9:678. doi: 10.3389/fneur.2018.00678. eCollection 2018. PMID 30174647
- [Background] Mutch WAC, El-Gabalawy R, Ryner L, Puig J, Essig M, Kilborn K, Fidler K, Graham MR. Brain BOLD MRI O2 and CO2 stress testing: implications for perioperative neurocognitive disorder following surgery. Crit Care. 2020 Mar 4;24(1):76. doi: 10.1186/s13054-020-2800-3. PMID 32131878
- [Background] Mutch WAC, El-Gabalawy RM, Graham MR. Postoperative Delirium, Learning, and Anesthetic Neurotoxicity: Some Perspectives and Directions. Front Neurol. 2018 Mar 20;9:177. doi: 10.3389/fneur.2018.00177. eCollection 2018. PMID 29615969
- [Background] El-Gabalawy R, Patel R, Kilborn K, Blaney C, Hoban C, Ryner L, Funk D, Legaspi R, Fisher JA, Duffin J, Mikulis DJ, Mutch WAC. A Novel Stress-Diathesis Model to Predict Risk of Post-operative Delirium: Implications for Intra-operative Management. Front Aging Neurosci. 2017 Aug 18;9:274. doi: 10.3389/fnagi.2017.00274. eCollection 2017. PMID 28868035
- [Background] Mutch WAC, El-Gabalawy R. Anesthesia and postoperative delirium: the agent is a strawman - the problem is CO2. Can J Anaesth. 2017 Jun;64(6):678-680. doi: 10.1007/s12630-017-0859-3. Epub 2017 Mar 10. No abstract available. PMID 28283991
- [Background] Ellis MJ, Ryner LN, Sobczyk O, Fierstra J, Mikulis DJ, Fisher JA, Duffin J, Mutch WA. Neuroimaging Assessment of Cerebrovascular Reactivity in Concussion: Current Concepts, Methodological Considerations, and Review of the Literature. Front Neurol. 2016 Apr 29;7:61. doi: 10.3389/fneur.2016.00061. eCollection 2016. PMID 27199885